CLINICAL TRIAL: NCT06378047
Title: A Phase 1 Study of Irreversible Electroporation and Pembrolizumab Immunotherapy in Locally Advanced Pancreatic Cancer
Brief Title: Irreversible Electroporation & Pembro Immunotherapy in Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22325
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer; Locally Advanced Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pembrolizumab; Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IRE/Pembrolizumab (Experimental): Participants will undergo irreversible electroporation (IRE) using the NanoKnife system. About 1 week following IRE, study participants will receive a 200mg dose of pembrolizumab.
  Interventions: Drug: Pembrolizumab; Device: Irreversible Electroporation

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is an immunotherapy that will be administered via IV infusion.
  Other Names: Keytruda
Device: Irreversible Electroporation — Participants will undergo IRE as standard of care treatment.
  Other Names: NanoKnife

SUMMARY:
This study aims to determine the safety and tolerability of combining sequential therapy of Irreversible Electroporation (IRE) and Immunotherapy (IO) for patients with locally advanced unresectable pancreas cancer following first-line treatment with chemotherapy and ablative stereotactic magnetic resonance image-guided adaptive radiation therapy (A-SMART).

ELIGIBILITY:
Inclusion Criteria:

* Participant must consent to enrollment in the Moffitt Cancer Center (MCC) Total Cancer Care (TCC) Protocol for tissue and blood banking and must have their initial biopsy tissue available.
* Participant must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, biopsies when required, and other procedures.
* Histologically or cytologically confirmed PDAC meeting the AJCC 8th edition staging criteria of stage 3 disease.
* Tumor(s) is/are locally advanced and unresectable pursuant to NCCN guidelines.
* Participant must be age 18-74 years at diagnosis.
* Performance-status Eastern Cooperative Oncology Group (ECOG) of 0-1.
* Radiologically measurable disease per iRECIST version 1.1.
* Prior to TCC registration, participants must have no prior therapy for PDAC and fall under treatment NCCN pancreatic adenocarcinoma guides (v1.2022) for locally advanced disease. Before study consent, the participant must have had standard of care first-line therapy consisting of 12 weeks of FOLFIRINOX (at least 6 cycles), followed by 50 Gy of A-SMART, delivered in five 10-Gy fractions. Participant must show no evidence of disease progression after first-line treatment, based upon National Comprehensive Cancer Network (NCCN) guidelines.
* The maximum axial tumor dimension must be ≤3.5 cm after "first strike" standard of care treatment.
* Participants must have adequate organ and marrow function.
* Resolved acute effects of any prior therapy and/or grade ≤1 late toxicity according to CTCAE version 5.0.
* If a participant requires anticoagulation, treatment must be modified to enoxaparin.
* Negative serum pregnancy test if female participant is of child-bearing potential. At screening, all female participants of child-bearing age will undergo a urine pregnancy test. If urine test is positive or inconclusive, a serum test will be performed.
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. In addition, WOCBP must agree to continue using adequate contraception for 4 months after pembrolizumab administration. If a woman is breastfeeding, she should stop study drug.
* Patients must be eligible for standard of care (SoC) NanoKnife therapy.

Exclusion Criteria:

* Clinical evidence of Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE), prior history of Cerebral Vascular Accident (CVA), or history of Transient Ischemic Attack (TIA) within 12 months or other known TE event present during the screening period.
* Clinically significant (i.e., active) cardiovascular disease: myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), serious cardiac arrhythmia requiring medication.
* Participants who have implanted cardiac pacemakers, defibrillators, or implanted devices with bare metal parts in the thoracic cavity, abdomen, and/or retroperitoneum.
* Currently receiving treatment with medication that has a known risk to prolong the QT interval or to induce Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting study treatment.
* Participant has other concurrent severe and/or uncontrolled medical conditions that would, in the Investigator's judgment, contraindicate patient participation in the clinical study.
* Contraindication to heparin as per institutional guidelines.
* Another primary cancer within the last 3 years requiring systemic therapy.
* Participant has had major surgery within 14 days prior to starting study treatment or has not recovered from major side effects.
* Participant is currently receiving increasing or chronic treatment (>5 days) with corticosteroids or another immunosuppressive agent within 2 weeks of study participation or has an active autoimmune disease that might deteriorate when receiving an immunostimulatory agent.
* Participant is being treated at start of study treatment with any of the following drugs: a. Drugs known to be strong or moderate inhibitors or inducers of isoenzyme cytochrome P450 3A4 (CYP3A4), including herbal medications. b. Drugs with a known risk of inducing Torsades de Pointes. Note: The patient must have discontinued strong inducers for at least 1 week and must have discontinued strong inhibitors before the treatment is initiated. Switching to a different medication prior to starting study treatment is allowed.
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Known prior severe hypersensitivity to investigational product, hyaluronidase, or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE version 5 grade ≥ 3).
* Participant has a medically documented poorly controlled psychiatric disorder(s), alcohol abuse, or drug abuse as defined according to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-V).
* Gastrointestinal arteriovenous malformations.
* Local gastrointestinal organ (e.g., stomach, duodenum) invasion by tumor.
* Participant is unable to undergo magnetic resonance imaging (MRI) due to incompatible implanted device, body habitus, and/or phobia unamenable to anxiolytic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Up to 90 days
  The number of participants who experience a high-grade (grade 3-5) adverse events based on NCI common terminology criteria for adverse events (CTCAE) version 5 related to treatment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months
  PFS is defined as the time from date of diagnosis to the time of first documented tumor progression or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 24 months
  OS is defined as the time from date of diagnosis to the time of death due to any cause.
Objective Response Rate (ORR) | Up to 24 months
  ORR is defined as the proportion of patients with either a partial or complete response according to iRECIST version 1.1 guidelines, measured from date of diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mokenge Malafa, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States